CLINICAL TRIAL: NCT02861820
Title: Functional Connectivity Changes During Early Recovery as a Marker for Relapse
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2016-24183; 1R01DA038984-01A1 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Substance Use Disorder
Keywords: fMRI; brain networks; biomarker; relapse; stimulants
MeSH Terms: conditions — Substance-Related Disorders; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Substance Use Disorder (SUD): Participants in the SUD group will:
  * Complete a diagnostic screening interview at baseline.
  * Complete questionnaires and computer tasks at baseline, 1 month and 2 month time points.
  * Complete MRI brain imaging data collection at the baseline, 1 month and 2 month time points.
  * Complete 9 follow-up phone calls to assess for relapse.
  Interventions: Device: MRI: Brain Imaging Data Collection
- Healthy Control (HC): Participants in the HC group will:
  * Complete a diagnostic screening interview at baseline.
  * Complete questionnaires and computer tasks at baseline and 2 month time points.
  * Complete MRI brain imaging data collection at the baseline and 2 month time points.
  Interventions: Device: MRI: Brain Imaging Data Collection

INTERVENTIONS:
Device: MRI: Brain Imaging Data Collection — This study has no intervention, it is observational. The investigator will collect brain imaging data and behavioral assessments.

SUMMARY:
The study purpose is to examine whether there are structural or functional differences in the brains of individuals who use cocaine or amphetamines as opposed to control participants who have never used cocaine or amphetamines. More specifically, it will allow the investigator to see how the brain changes once people get sober and how those changes relate to successful recovery. This study will allow the investigator to examine the interaction between cocaine/amphetamines and impulsivity (meaning to act on impulse rather than thought). Results from this study will inform new biologically-based interventions to compliment existing treatment programs, in the hope of leading the field in a new direction.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 but no more than 45 years old at the time of consent.
* Able to provide written consent and comply with study procedures.

Exclusion Criteria:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness for more than 30 minutes, seizures, HIV).
* Any contraindications to MRI scanning (i.e. metal implants, pacemakers, etc.).
* Intellectual developmental disorder as defined in the DSM-V. Participant may have a diagnosis of an Axis I disorder (i.e. anxiety disorders, mood disorders, eating disorders, psychotic disorders), but it must be considered stable.
* Actively suicidal.
* Positive screen for alcohol and/or drugs. Participants who screen positive for drugs and/or alcohol may return at a later date to screen for the study again.
* Evidence for Wernicke-Korsakoff syndrome.
* Healthy Controls may never have had any form of substance use disorder other than caffeine or nicotine. Nicotine use will be recorded but will not be an exclusion criterion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult individuals with Substance Use Disorder
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Brain connectivity | Change from Baseline, to 2 months
  3T MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin O Lim, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
As requested

DOCUMENTS (1):
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT02861820/ICF_000.pdf